CLINICAL TRIAL: NCT04530968
Title: Metabolic Abnormalities and Intestinal Microecology in Patients With Chronic Disorders of Consciousness
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: microbiome and metabolomic
Record Dates: First submitted 2020-07-29; First posted 2020-08-28 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2020-07

CONDITIONS: Disorder of Consciousness
Keywords: Disorder of Consciousness; microbiome; metabolomics
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma for metabolites and lipids；Fecal samples for microbiome and metabolites.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Emerged from Minimally Conscious State (EMCS): Emerged from Minimally Conscious State (EMCS): recovery of functional object uses or communication from chronic
  Interventions: Other: No intervention
- Minimally conscious state (MCS): Minimally conscious state (MCS): have reproducible signs of awareness and exhibit fluctuations in consciousness
  Interventions: Other: No intervention
- Vegetative state (VS): Vegetative state (VS): can open their eyes and preserve sleep-wake cycles, but unaware of themselves and their surroundings
  Interventions: Other: No intervention
- Healthy controls (HCs): Healthy controls (HCs)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Following severe traumatic brain injury, patients may remain unconscious for many years. It is the intestinal microbiome and metabolomics analysis comparing differentially intestinal microflora and metabolites between patients with chronic disorder of consciousness and controls so far. The investigators have mature data analysis technology. The obtained results provide new insight into understanding the molecular mechanisms underlying the chronic disorder of consciousness

DETAILED DESCRIPTION:
Objective:To determine differences in metabolic profiles and Intestinal microbial abundance among healthy human individuals and patients in a vegetative state (VS) and minimally conscious state (MCS) and to identify metabolites in human plasma that can accurately distinguish VS patients from MCS patients.

Method: Plasma samples and fecal sample were obtained from patients with chronic disorder of consciousness, and healthy volunteers. A comprehensive metabolic profile was obtained with targeted metabolomics analysis and untargeted and targeted lipidomics analysis, as well as intestinal microbial abundance from 16S rRNA gene amplicon sequencing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 18 to 80 years old;
2. Patients had a history of severe Traumatic brain injury (TBI);
3. Patients had awakened from a coma (indicating preserved sleep-wake cycles), including vegetative state and minimally consciousness state;
4. Patients stay unconscious for more than 1 month.

Exclusion Criteria:

1. Patients with disorders of consciousness caused by other inducements;
2. Other neurological or psychiatric conditions prior to the current brain injury;
3. Persistent seizure-like activity, inhibition or seizure inhibition;
4. The patients had taken a sedative barbiturate neuroleptics or antidepressants within one month;
5. The clinical state is unstable, and there are signs of spontaneous recovery or deterioration within 1 week;
6. The patients have taken gastrointestinal motility drugs or other drugs affecting gastrointestinal motility in the past month;
7. Had taken antibiotics and probiotics in the past month;
8. Patients with intestinal diseases such as colon cancer, ulcerative colitis or crohn's disease;
9. Patients with acute infectious diseases or liver dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic disorder of consciousness were recruited at the rehabilitation units of Hangzhou Hospital of Zhejiang Armed Police Corps, China and Hangzhou Mingzhou Brain Rehabilitation Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
metabolic profiling and Intestinal microbial spectrum | 1 month
  A comprehensive metabolic profile from plasma was obtained with targeted metabolomics analysis and untargeted and targeted lipidomics analysis; intestinal microbial spectrum was obetained from fecal by16S rRNA gene sequencing among HCs, EMCS, MCS and VS groups.

SECONDARY OUTCOMES:
Coma Recovery Scale-Revised(CRS-R) | 30 minutes before samples collection
  Coma Recovery Scale-Revised (CRS-R) score was used to quantify the severity, which consists of 23 hierarchically arranged items that comprise six subscales addressing auditory, visual, motor, oromotor/verbal, communication, and arousal processes. The lowest item on each subscale represents reflexive activity, whereas the highest items represent cognitively mediated behaviors In total, The lowest mark on the scale is 0 and the highest mark is 23. To a certain extent, the higher the score is, the better the level of consciousness is, whereas the lower the level of consciousness is.
Glasgow Outcome Scale (GOS) | 6 months
  A GOS value of <3 was considered as a bad recovery, while a GOS value of ≥3 was considered as a good recovery.
Indicators of brain connectivity by EEG | On the same day as collecting the samples
  Phase locking value (PLV)

CONTACTS AND LOCATIONS:
Locations (1):
- SCIEX QTRAP 5500 liquid chromatograph / triple quadrupole mass spectrometer., Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No